CLINICAL TRIAL: NCT01797003
Title: Time-dependent Functional Results Following HTO. Closing Wedge vs Opening Wedge Technique.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Tor Kjetil Nerhus, Consultant Orthopaedic surgeon, Vestre Viken Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKN-003
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; osteotomy; closing; opening; wedge; kne; tibia
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opening wedge HTO (Active Comparator): Opening wedge high tibial osteotomy using Puddu plate
  Interventions: Other: High tibial osteotomy
- Closing wedge HTO (Active Comparator): Closing wedge high tibial osteotomy using cramp fixation
  Interventions: Other: High tibial osteotomy

INTERVENTIONS:
Other: High tibial osteotomy

SUMMARY:
Prospective randomized study. Compare two techniques for high tibial osteotomy (HTO) for treatment of medial knee osteoarthritis.

Opening wedge osteotomy using Puddu plate vs Closing wedge osteotomy using cramp fixation. We will compare functional results and patient satisfaction with repetitive evaluations from preoperatively to 2 years postoperatively.

DETAILED DESCRIPTION:
Determination of the time course of patient-relevant functional outcome and the time course of Range of Motion (ROM) following HTO. Comparison of the Opening wedge and Closing wedge methods.

Time-dependent improvement in functional outcome following High tibial Osteotomy. Medial opening wedge vs Lateral closing wedge. A two-year prospective randomized study involving 70 patients.

In a prospective randomized study, we plan to include 70 patients aged 30-60 years operated with valgus high tibial osteotomy. 2 groups: 35 opening wedge, and 35 closing wedge osteotomies. Data are collected by independent investigators (physiotherapists) preoperatively and at 3 months, 6 months, 1 year, and 2 years postoperatively. Knee injury and Osteoarthritis Outcome Score (KOOS) and ROM are determined at all follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Medial osteoarthritis in the knee (x-ray and arthroscopy)
* Pain in medial compartment of the knee
* Correction angle of 5 degrees or more

Exclusion Criteria:

* Former or active infection in the knee
* Rheumatoid arthritis or other similar disease
* Cancer
* Neurological disease
* Kidney disease or metabolic disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2007-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Kne injury and Osteoarthritis Outcome Score (KOOS) | 2 years postoperataively
  The change in KOOS score are followed at several time points the first 2 years. Patients will be evaluated with KOOS, 3 months, 6 months, 1 year and 2 years postoperatively.

SECONDARY OUTCOMES:
Range of motion (ROM) | 2 years postoperatively
  The change in ROM are followed at several time points the first 2 years. ROM will be measured 3 months, 6 months, 1 year and 2 years postoperatively.

OTHER OUTCOMES:
Oxford knee score | 2 years
  The change in Oxford score are followed at several time points the first 2 years. Patients will be evaluated with Oxford knee score, 3 months, 6 months, 1 year and 2 years postoperatively.
Lysholm score | 2 years postoperatively
  The change in Lysholm score are followed at several time points the first 2 years. Patients will be evaluated with Lysholm, 3 months, 6 months, 1 year and 2 years postoperatively.
UCLA activity scale | 2 years postoperatively
  The change in UCLA scale are followed at several time points the first 2 years. Patients will be evaluated with UCLA activity scale, 3 months, 6 months, 1 year and 2 years postoperatively.
Tegner Activity Score | 2 years postoperatively
  The change in Tegner score are followed at several time points the first 2 years. Patients will be evaluated with Tegner score, 3 months, 6 months, 1 year and 2 years postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Kjetil Nerhus, MD, Principal Investigator — Consultant orthopaedic surgeon
Locations (1):
- Martina Hansens Hospital, Oslo, Norway